CLINICAL TRIAL: NCT02638597
Title: Gemfibrozil for Nicotine Smoking Cessation
Acronym: GEMNIC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Madhukar H. Trivedi, MD, Madhukar H. Trivedi, MD, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU 072014-088
Record Dates: First submitted 2015-12-18; First posted 2015-12-23 (Estimated); Results first posted 2019-02-01 (Actual); Last update posted 2019-02-01 (Actual); Status verified 2019-01

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — Gemfibrozil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gemfibrozil (Experimental): Participants in this arm will receive smoking cessation counseling and will be provided gemfibrozil 600 mg twice daily by mouth for 9 weeks, starting one week prior to target quit date and ending with study completion
  Interventions: Drug: Gemfibrozil; Behavioral: smoking cessation counseling
- Waitlist (Other): Participants in this arm will receive the smoking cessation counseling but will not receive medication. After completing the trial without medication, participants who continue to smoke and have a desire to quit may choose to enter the gemfibrozil arm.
  Interventions: Behavioral: smoking cessation counseling

INTERVENTIONS:
Drug: Gemfibrozil — FDA Approved Drug(s)/Biologic(s) (study use is not an FDA-approved use)
  Other Names: Lopid
  Arms: Gemfibrozil
Behavioral: smoking cessation counseling — smoking cessation counseling

SUMMARY:
This project will test whether gemfibrozil, a well-studied medication for high cholesterol, will help people stop smoking nicotine cigarette smoking. The study will also test whether gemfibrozil decrease cravings for cigarette and the desire to smoke.

DETAILED DESCRIPTION:
This is a pilot clinical trial examining the feasibility and efficacy of gemfibrozil treatment for smoking cessation. Adults with a desire to quit nicotine cigarette smoking will be recruited. Eligible participants will be randomly divided into two groups: those who receive gemfibrozil and waitlist controls. Screening will be conducted with a brief phone screen followed by a longer screening visit for those who qualify. During the screening visit, all study participants will provide demographic information and will be interviewed regarding smoking history. Procedures performed during the screening visit include a blood draw, urine pregnancy test, physical exam, clinical psychiatric interview, and measurement of exhaled carbon monoxide (CO). At baseline, participants will complete the Heavy Smoking Index (HSI) and the Brief Questionnaire of Smoking Urges (QSU-Brief). Participants will also complete the Quick Inventory of Depressive Symptoms-Self Rated (QIDS-SR) to assess symptoms of depression and changes in mood associated with smoking cessation will be assessed with the Concise Associated Symptoms Tracking (CAST) scale . Participants will work with the research clinician to set a target quit date within one week of the baseline session, and all participants will be provided written materials with guidance for smoking cessation as part of a smoking cessation counseling session. All participants will attend visits at the research clinic at 3 days and 4 weeks from target quit date to assess safety, adherence, and smoking status; participants will also receive additional smoking cessation counseling. Smoking status will be determined with exhaled breath CO and a single item questionnaire regarding the number of cigarettes smoked since target quit date and symptoms of depression and mood changes will again be measured. Medication side effects will be quantified using the Frequency, Intensity, and Burden of Side Effects Rating (FIBSER) scale. The final study visit will occur at 8 weeks after target quit date for completion of the HSI, QIDS-SR, CAST, FIBSER, exhaled breath CO, QSU-Brief, and smoking self-report.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-64 years
* Meet DSM-5 criteria for tobacco use disorder based on cigarette use
* Desire to quit smoking
* Able to complete assessments and interview in English

Exclusion Criteria:

* Psychiatric co-morbidity posing safety risk, including current suicidality or psychosis as assessed on clinical interview
* Concurrent use of a statin medication (HMG-CoA reductase inhibitor),anticoagulant, or repaglinide
* Concurrent use of any FDA-approved medication for smoking cessation
* Use of any form of tobacco or nicotine (including vaporizer) other than cigarette smoking
* Any DSM-5 substance use disorder other than nicotine use disorder
* History of intolerance to any fibrate medication
* History of gallbladder disease and cholestectomy has not been performed
* Baseline liver function tests > twice the upper limit of normal
* Severe impairment of renal function (baseline serum creatinine ≥ 2 mg/dL)
* Currently pregnant or nursing

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2015-02; Primary Completion 2016-12-23 (Actual); Study Completion 2016-12-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Madhukar Trivedi, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- Parkland Memorial Hospital, Dallas, Texas, United States

REFERENCES:
- [Background] Rush AJ, Trivedi MH, Ibrahim HM, Carmody TJ, Arnow B, Klein DN, Markowitz JC, Ninan PT, Kornstein S, Manber R, Thase ME, Kocsis JH, Keller MB. The 16-Item Quick Inventory of Depressive Symptomatology (QIDS), clinician rating (QIDS-C), and self-report (QIDS-SR): a psychometric evaluation in patients with chronic major depression. Biol Psychiatry. 2003 Sep 1;54(5):573-83. doi: 10.1016/s0006-3223(02)01866-8. PMID 12946886
- [Background] Trivedi MH, Wisniewski SR, Morris DW, Fava M, Kurian BT, Gollan JK, Nierenberg AA, Warden D, Gaynes BN, Luther JF, Rush AJ. Concise Associated Symptoms Tracking scale: a brief self-report and clinician rating of symptoms associated with suicidality. J Clin Psychiatry. 2011 Jun;72(6):765-74. doi: 10.4088/JCP.11m06840. PMID 21733477
- [Background] Wisniewski SR, Rush AJ, Balasubramani GK, Trivedi MH, Nierenberg AA; STARD Investigators. Self-rated global measure of the frequency, intensity, and burden of side effects. J Psychiatr Pract. 2006 Mar;12(2):71-9. doi: 10.1097/00131746-200603000-00002. PMID 16728903

RESULTS

PARTICIPANT FLOW:
Groups:
- Waitlist: Participants placed on waitlist for medication, otherwise completed study procedures
- Gemfibrozil: Received gemfibrozil tablets
Period: Overall Study
Arm/Group | Waitlist | Gemfibrozil
Started | 8 | 8
Completed | 4 | 3
Not Completed | 4 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Waitlist | Gemfibrozil | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 8 | 16
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 25.25 (14.12) | 37.50 (22.02) | 31.38 (18.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 2 | 2 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8 | 8 | 16

OUTCOME MEASURES:

1. Primary Outcome: Exhaled Carbon Monoxide (CO)
Description: Exhaled carbon monoxide change from baseline to last available visit.
Time Frame: 8 weeks after target quit date
Measure: Mean (Standard Deviation); unit: Parts p/million
Arm/Group | Gemfibrozil | Waitlist
Number analyzed (Participants) | 8 | 8
Parts p/million | 10.88 (12.63) | 21.63 (22.04)

2. Secondary Outcome: Heaviness of Smoking Index
Description: The outcome measure was Heaviness of Smoking Index at exit. The Heaviness of Smoking Index is a two-item scale, with scores on each item rated on a 1-4 likert scale. The total score of the measure ranges from 2-8, with higher scores indicating worse outcome.
Time Frame: 8 weeks after target quit date
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Waitlist | Gemfibrozil
Number analyzed (Participants) | 8 | 8
score on a scale | 1.25 (1.04) | 1.63 (1.30)

ADVERSE EVENTS:
Arm/Group | Gemfibrozil | Waitlist
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 1/8 | 1/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gemfibrozil (N=8) | Waitlist (N=8)
Arm bruising (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Arm bruising as a result of study-related blood draw.
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) — Ended up being gallbladder disease.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes